CLINICAL TRIAL: NCT06145230
Title: A Cross-sectional Survey of Symptomatic Characteristics, Family History and Pathologic Features of Colorectal Cancer Patients in Different Age Groups
Brief Title: A Cross-sectional Survey of Colorectal Cancer Patients in Different Age Groups
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wang Guiyu (Other)
Responsible Party: Sponsor-Investigator, Wang Guiyu, Director of the Department of Colorectal Cancer Surgery, The Second Affiliated Hospital of Harbin Medical University
Organization: The Second Affiliated Hospital of Harbin Medical University (Other)
Other Study IDs: 2ndHarbinMUSUV
Record Dates: First submitted 2023-10-09; First posted 2023-11-24 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Age Problem
Keywords: Colorectal caner; Age group; Family history; Symptomatic characteristics; Pathologic features
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Under 60 group: Colorectal cancer paitents aged under 60 years old ( do not include 60 years old)
- 60-69 group: Colorectal cancer paitents aged 60-69 years old
- 70-79 group: Colorectal cancer paitents aged 70-79 years old
- 80 and over group: Colorectal cancer paitents aged 80 and over 80 years old

INTERVENTIONS:
Other:

SUMMARY:
This study will help to determine the main clinical symptom differences between patients of different ages, discover the family genetic predisposition of patients of different ages, and obtain the differences in pathological characteristics of patients of different ages, so as to provide help and basis for more accurate and earlier prevention and treatment of colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is one of the common and highly prevalent malignant tumors of the gastrointestinal system. Previous studies have found that there may be some differences in disease characteristics and prognosis of colorectal cancer patients at different ages, such as patients with early-onset colorectal cancer (age <50 years) tend to have a worse prognosis than patients with late-onset colorectal cancer (age ≥50 years). However, existing studies on the characteristics of colorectal cancer patients at different ages are not well studied to answer the differences between these patients and develop targeted diagnostic and treatment strategies. Cross-sectional survey research, which uses survey research to collect data on a characteristic group over a certain period of time and statistically analyzes the data to obtain the characteristics of a certain disease or a certain treatment strategy, is a more mature approach that is particularly suitable for the questions that need to be answered in this study. Investigators found that no similar studies have been registered and conducted by searching the official websites of the China Clinical Research Registry and Clinical Trial, and there is a lack of research data on the Chinese population. Therefore, investigators believe there is an urgent need for a cross-sectional survey to study the symptomatic characteristics, family history, and pathologic features of colorectal cancer patients. This study will help to determine the main clinical symptom differences between patients of different ages, discover the family genetic predisposition of patients of different ages, and obtain the differences in pathological characteristics of patients of different ages, so as to provide help and basis for more accurate and earlier prevention and treatment of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older with a pathologic diagnosis of colorectal cancer;
2. Undergoing surgical treatment of the primary lesion;
3. Voluntary participation of patients.

Exclusion Criteria:

1. Do not agree to participate in the survey or withdraw informed consent
2. Patients did not receive surgical treatment or did not undergo pathologic examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation of gender identity
Study Population: Colorectal cancer patients in different age groups
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of clinical symptoms | 2023.12-2024.10
  Comparison of the characteristics of clinical symptoms in patients of different ages;
Family history | 2023.12-2024.10
  Comparison of the probability of having a family history in patients of different age stages;
Pathological characteristics | 2023.12-2024.10
  Comparison of pathological characteristics of patients at different age stages;

SECONDARY OUTCOMES:
Risk factors | 2024.09-2024.10
  Analysis of risk factors for stage progression in colorectal cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Ye Tian, Prof., Study Chair — Second Affiliated Hospital of Harbin Medical University Ethics Committee
Locations (1):
- the 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China